CLINICAL TRIAL: NCT04054830
Title: Steroids and/ or Non-steroidal Anti-inflammatory Drugs in the Postoperative Regime After Trabeculectomy. An Investigator-initiated Randomized Study (The SNAP Study)
Brief Title: Steroids and/ or Non-steroidal Anti-inflammatory Drugs in the Postoperative Regime After Trabeculectomy.
Acronym: SNAP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Afrouz Ahmadzadeh, MD, PhD-student, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EudraCT nr.: 2018-001855-10
Record Dates: First submitted 2019-08-09; First posted 2019-08-13 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Glaucoma
Keywords: Trabeculectomy; NSAID; Steroid; Anti-Inflammatory Agents; Anti-Inflammatory Agents, Non-Steroidal; Eye Diseases
MeSH Terms: conditions — Glaucoma; Eye Diseases | interventions — halofantrine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Topical, preservative-free NSAID (Experimental): Topical medication are to be used 6 times daily for the 2 first weeks, tapering to 4 drops per day for the next 4 weeks. Depending on the clinical condition of the eye, the topical anti-inflammatory treatment will be reduced with 1 daily drop per week.
  Interventions: Drug: Voltaren Ophtha 1 mg/ml, GSK
- Topical, preservative-free steroid (Active Comparator): Topical medication are to be used 6 times daily for the 2 first weeks, tapering to 4 drops per day for the next 4 weeks. Depending on the clinical condition of the eye, the topical anti-inflammatory treatment will be reduced with 1 daily drop per week.
  Interventions: Drug: Monopex 1 mg/ml, Théa
- Topical, preservative-free NSAID (Voltaren Ophtha 1 mg/ml, GSK (Experimental): Topical medication are to be used 6 times daily for the 2 first weeks, tapering to 4 drops per day for the next 4 weeks. Depending on the clinical condition of the eye, the topical anti-inflammatory treatment will be reduced with 1 daily drop per wee
  Interventions: Drug: Voltaren Ophtha 1 mg/ml, GSK; Drug: Monopex 1 mg/ml, Théa

INTERVENTIONS:
Drug: Voltaren Ophtha 1 mg/ml, GSK — Voltaren Ophtha 1 mg/ml, eye drops used 6 times daily for the 2 first weeks, tapering to 4 drops per day for the next 4 weeks. Depending on the clinical condition of the eye, the topical anti-inflammatory treatment will be reduced with 1 daily drop per week.
  Arms: Topical, preservative-free NSAID; Topical, preservative-free NSAID (Voltaren Ophtha 1 mg/ml, GSK
Drug: Monopex 1 mg/ml, Théa — Monopex 1 mg/ml, eye drops used 6 times daily for the 2 first weeks, tapering to 4 drops per day for the next 4 weeks. Depending on the clinical condition of the eye, the topical anti-inflammatory treatment will be reduced with 1 daily drop per week.
  Arms: Topical, preservative-free NSAID (Voltaren Ophtha 1 mg/ml, GSK; Topical, preservative-free steroid

SUMMARY:
PURPOSE:

Glaucoma is the leading cause of non-curable blindness globally. Patients with glaucoma will get a gradual narrowing of the visual fields caused by compression at the optic nerve head due to increased intraocular pressure. Thus the main preventive strategy is to reduce intraocular pressure, initially by eye drops and/or laser treatment but in some patients surgery is warranted. The surgical procedure (trabeculectomy) most widely performed worldwide creates a path from the anterior chamber to the subconjunctival space and thereby lowers the IOP by producing a more efficient drainage of the aqueous humour. Surgical success depends upon controlling post-operative inflammation to ensure a functional drainage. The purpose of this blinded, randomized study is to investigate which anti-inflammatory treatment provides better long-term control of intra-ocular pressure (IOP) following glaucoma surgery (trabeculectomy) by comparing topical NSAIDs to topical steroids. Additionally, we want to explore the mechanisms behind the pathophysiology of glaucoma by evaluating retinal and optic nerve head perfusion before and after IOP lowering surgery. The primary outcome is the intraocular pressure 12 months after surgery measured by applanation tonometry.

MAIN HYPOTHESIS:

* NSAIDs and steroids are equally effective in assuring long-term filtering function and controlling IOP after trabeculectomy but may be associated with different risk profiles and bleb morphology
* Patients with lower post-operative IOP demonstrate less progression of visual field loss
* Trabeculectomy lowers IOP and provides better microcirculation in and oxygenation of inner retinal layers (i.e. ganglion cell layer) and the optic nerve head

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary open-angle glaucoma (POAG), pseudoexfoliation syndrome (PEX), pigment dispersion syndrome (PDS) or ocular hypertension
* >50 years
* Women must be postmenopausal. Women are asked if they have menstruated within the preceding 12 months
* Scheduled to undergo trabeculectomy surgery at the Department of Ophthalmology at Rigshospitalet-Glostrup, Denmark
* Informed consent to participation and ability to comply with study procedures

Exclusion Criteria:

* Known allergy to any of the contents of the pharmaceuticals (active and in-active ingredients) used in the study
* Prior intraocular surgery, except from cataract surgery. If cataract surgery has been performed, it should at least be 6 months prior to surgery
* Medical history of anterior segment dysgenesis, inflammatory/uveitic glaucoma, angle closure glaucoma, neovascular glaucoma and traumatic glaucoma
* Steroid responders
* Pregnancy
* Fertile women, i.e. women who are not menopausal and women who breastfeed
* Patients in systemic treatment with steroid or NSAID

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure (IOP) | 12 months
  Postoperative intraocular pressure (IOP) by applanation tonometry

SECONDARY OUTCOMES:
Best corrected visual acuity | 12 months, 24 months
  Postoperative best corrected visual acuity in logarithm to the minimal angle of resolution (logMAR)
Visual field | 12 months, 24 months
  Postoperative changes in visual field by octopus autoperimetry. (MD)
Optical nerve damage | 12 months, 24 months
  Optical nerve damage, assessed by measuring retinal nerve fiber layer (RNFL) by peripapillary optical coherence tomography (OCT)
Surgical success | 12 months, 24 months
  The definition of surgical success criteria is dependent on the the severity of visual field defect (MD, mean deviation of visual sensitivity compared to those expected from the age-matched normative database) glaucoma diagnosis and achievement of target pressure without the use of medication (complete success) or with the use of glaucoma medication (qualified success)
  * Ocular hypertension, target <25 mmHg
  * MD < 6 dB, target < 21 mmHg
  * MD 6 dB - 12 dB, target <18 mmHg
  * MD > 12 dB, target < 15 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Daniella Bach-Holm, MD, Ph.D., Principal Investigator — Dpt. of Ophthalmology, Rigshospitalet-Glostrup
Locations (1):
- Department of Ophthalmology, Glostrup Municipality, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ahmadzadeh A, Schmidt BS, Bach-Holm D, Kessel L. Early Inflammation Control After Trabeculectomy by Steroid and Non-steroidal Eye Drops: A Randomized Controlled Trial. Ophthalmol Ther. 2023 Apr;12(2):969-984. doi: 10.1007/s40123-022-00636-2. Epub 2023 Jan 5. PMID 36602718